CLINICAL TRIAL: NCT06346730
Title: The Effect of Virtual Reality Application on Anxiety and Patient Satisfaction During Intrauterine Insemination (IUI): Randomized Controlled Study
Brief Title: The Effect of Virtual Reality Application on Anxiety and Patient Satisfaction During Intrauterine Insemination (IUI)
Acronym: (IUI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ayşe Sevim AKBAY KISA, Investigator, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 142-18
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Virtual Reality; Anxiety; Patient Satisfaction; Intrauterine Insemination (IUI)
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: The sample will divide into intervention and control groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality glasses to intervention group (Experimental): Virtual reality glasses to intervention group, randomized pretest-posttest
  Interventions: Device: Virtual reality glasses to intervention group
- control (No Intervention): Non-intervention

INTERVENTIONS:
Device: Virtual reality glasses to intervention group — experimental and control ,a randomized pretest-posttest study to examine
  Arms: Virtual reality glasses to intervention group

SUMMARY:
This study will conduct as a randomized pretest-posttest study to examine the effect of virtual reality glasses (VRG) application during the IUI procedure on anxiety and patient satisfaction. The population of the research will consist of women who were treated with assisted reproductive techniques and underwent IUI at the infertility polyclinic of Ministry of Health Adana City Training and Research Hospital between May and December 2024 and who meet the research criteria. The research sample was calculated as a total of 90 people (at least 45 people in each group) using the power program. Data; Personal Information Form, Visual Assessment Scale (VAS), State Trait Anxiety Inventory (STAI) and Patient's Perception of Nursing Care Scale will be collected from women who agree to participate in the research. Virtual reality glasses will be applied to the intervention group.

DETAILED DESCRIPTION:
This study will conduct as a randomized pretest-posttest study to examine the effect of virtual reality glasses (VRG) application during the IUI procedure on anxiety and patient satisfaction. The population of the research will consist of women who were treated with assisted reproductive techniques and underwent IUI at the infertility polyclinic of Ministry of Health Adana City Training and Research Hospital between May and December 2024 and who meet the research criteria. The research sample was calculated as a total of 90 people (at least 45 people in each group) using the power program. Data; Personal Information Form, Visual Assessment Scale (VAS), State Trait Anxiety Inventory (STAI) and Patient's Perception of Nursing Care Scale will be collected from women who agree to participate in the research. These scales will be applied to both groups before and after Intrauterine Insemination (IUI).

Virtual reality glasses will be applied to the intervention group during intrauterine insemination (IUI).

Keywords: Virtual reality, anxiety, patient satisfaction, Intrauterine Insemination (IUI)

ELIGIBILITY:
Inclusion Criteria:

* 18-45 age group
* Primary infertile,
* Able to speak and understand Turkish,
* Are cognitive, effective and have no problems preventing communication,
* Having no psychiatric problems,
* Not diagnosed with epilepsy (due to the possibility of virtual reality (VR) glasses triggering epileptic seizures),
* Women who volunteer to participate in the study will be recruited.

Exclusion Criteria:

* Having a psychiatric problem,
* Diagnosed with epilepsy
* Those who want to leave the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory (STAI) | The research period for a participant takes approximately 30 minute
  State Trait Anxiety Inventory (STAI) was designed to identify individuals' persistent anxiety and the level of anxiety felt towards the situation they are in. A total score between 20 and 80 can be obtained from both scales. Measuring ranges; 20-39 points are considered mild, 40-59 points are considered moderate, 60-79 points are considered severe anxiety, and 80 points are considered panic.
Patient's Perception of Nursing Care Scale | The research period for a participant takes approximately 30 minute
  The Anxiety Inventory was designed to identify individuals' constant anxiety and the level of anxiety they feel about their current situation. A minimum of 15 and a maximum of 75 points can be obtained from the scale. An increase in the total score obtained from the scale indicates that the patient is satisfied with the nursing care.

CONTACTS AND LOCATIONS:
Overall Officials: Evşen ÇU NAZİK, professor, Study Chair — Cukurova University; Ayşe Sevim SU Akbay Kısa, Ph.D, Study Chair — Suleyman Demirel University; Ebru Var, Study Chair — Adana City Training and Research Hospital; Sefa ARLIER, professor, Study Chair — Adana City Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No